CLINICAL TRIAL: NCT00646503
Title: A Single Arm, Multicenter, Open-label, 52-week, the Omnibus Extension Study to Evaluate the Safety and Efficacy of Telbivudine in the Fifth Year of Treatment in Chinese Patients With Compensated Chronic Hepatitis B and Are HBV DNA PCR Negative at the End of Year 4 Treatment
Brief Title: Prospective Exploratory Study to Evaluate the Safety and Efficacy of Telbivudine in the Fifth Year of Treatment in Chinese Patients With Compensated Chronic Hepatitis B
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLDT600ACN04
Record Dates: First submitted 2008-03-26; First posted 2008-03-28 (Estimated); Last update posted 2017-06-22 (Actual); Status verified 2017-06

CONDITIONS: Hepatitis B, Chronic
Keywords: Hepatitis B, Chronic; Telbivudine; Polymerase Chain reaction
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Telbivudine

ARMS (1):
- 1 (Experimental): 600 mg/day, oral telbivudine for 52 weeks
  Interventions: Drug: Telbivudine

INTERVENTIONS:
Drug: Telbivudine — 600 mg/day, oral telbivudine for 52 weeks
  Other Names: SEBIVO; TYZEKA

SUMMARY:
This study will explore efficacy and safety of Telbivudine in the fifth year of treatment.

ELIGIBILITY:
Inclusion criteria

* Patient completed Omnibus study and will be available to immediately rollover into this study without discontinuation of study drug.
* Patient was not discontinued from the previous Omnibus study.
* Male or female, adult patients with CHB (HBeAg positive or HBeAg negative).
* Patient is willing and able to provide written informed consent to participate in the study.
* HBV DNA PCR undetectable in recent 12 months.

Exclusion criteria

* Pregnant or breastfeeding, or has plan of pregnant during study period.
* Patient is co-infected with hepatitis C virus (HCV), hepatitis D virus (HDV), r HIV at screening visit.
* Patient needs any anti-HBV treatment combination (add-on therapy) or switch to other anti HBV treatment from Telbivudine at investigator's discretion.
* Patient has any laboratory value abnormality that physicians think he/she may not be suitable to continue the Telbivudine treatment.
* Patient has any clinically significant concurrent severe or unstable disease conditions that physicians think he/she may have any additional risk or not be suitable to participate the study.
* Patient has evidence of renal insufficiency defined as patient requiring dialysis or having an estimated creatinine clearance below 50mL/min, as estimated by the cockcroft-Gault formula.
* Patient is currently abusing alcohol or illicit drugs.
* Patient is enrolled or plans to enroll in another clinical trial of an investigational agent while participating in this study.
* All other treatments for hepatitis B, including commercially available treatments indicated for conditions other than chronic hepatitis B that are being investigated to treat or may have activity against HBV (e.g., ribavirin, famciclovir, ganciclovir, etc.)
* Prolonged use of systemic acyclovir or famciclovir defined as episodic treatment with these agents for periods exceeding 10 days every 3 months, or chronic suppressive therapy.
* Systemic immunomodulators of any type.
* Systemic corticosteroids ( topical and inhaled corticosteroids are permitted).
* Herbal medications known to cause hepatotoxicity (e.g., St. John's Wart, Kava, Jin Bu Huan, Yuzhitang, germander, chaparral, shark cartilage, mistletoe, slim 10, Lipokinetix, etc.).
* Patient has any of the following laboratory values:

  * Hemoglobin < 9 g/dL for menor <8 g/dL for women.
  * Total WBC <1,500/mm3
  * Absolute neutrophil count (ANC)<1,000/mm3
  * Platelet count <30,000/mm3
  * Serum albumin <2.5g/dL
  * Total bilirubin ≥4×ULN
  * Serum creatinine >1.5×ULN

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2008-03; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Proportion of patients experiencing serious adverse events (for all SAEs, and SAEs attributed to study drug). Proportion of patients experiencing adverse events, coded by body system ( all AEs, and AEs attributed to study drug). | At Baseline, Week 24 and Week 52

SECONDARY OUTCOMES:
For HBeAg-positive patients, Maintained Virologic Response, here defined as HBeAg loss and serum HBV DNA PCR negative (COBAS Amplicor PCR < 300 copies/ml) during the whole study period. | At Baseline, Week 24 and Week 52

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis
Locations (1):
- Novartis Investigative Site, Beijing, China

REFERENCES:
- [Result] Hou JL, Xu D, Shi G, Wan M, Goodman Z, Tan D, Xie Q, Chen C, Wei L, Niu J, Wang Q, Ren H, Wang Y, Jia J, Bao W, Dong Y, Trylesinski A, Naoumov NV. Long-Term Telbivudine Treatment Results in Resolution of Liver Inflammation and Fibrosis in Patients with Chronic Hepatitis B. Adv Ther. 2015 Aug;32(8):727-41. doi: 10.1007/s12325-015-0232-2. Epub 2015 Sep 2. PMID 26329749